CLINICAL TRIAL: NCT02411500
Title: A Randomized, Open Label, Four Period, Cross-Over Study to Evaluate the Pharmacokinetics of Single Doses of Various TRV734 Formulations in Healthy Male Subjects
Brief Title: A Pharmacokinetic, Safety and Tolerability Study in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP734-1003
Record Dates: First submitted 2015-03-04; First posted 2015-04-08 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Healthy; Male; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Formulation A (Experimental)
  Interventions: Drug: TRV734
- Formulation B (Experimental)
  Interventions: Drug: TRV734
- Formulation C (Experimental)
  Interventions: Drug: TRV734
- Formulation D (Experimental)
  Interventions: Drug: TRV734
- Formulation E (Experimental)
  Interventions: Drug: TRV734
- Formulation F (Experimental)
  Interventions: Drug: TRV734

INTERVENTIONS:
Drug: TRV734 — Subjects will be randomized to receive the oral TRV734 treatments on Days 1, 3, 5 and 7 in an open-label, 4-period, cross-over fashion. Days 2, 4, 6 and 8 are designated as washout days.

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics of various TRV734 formulations in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician or trained qualified designee
* Males: 18 - 55 years inclusive at screening
* Capable of giving written informed consent

Exclusion Criteria:

* Clinically significant conditions or history of fainting or syncope
* Medical or psychiatric illness that could interfere with the completion of treatment and follow up
* Major surgery within 4-weeks of screening
* Known difficulty with obtaining intravenous access
* History of sensitivity to the study medication, or intolerance to opioids, or a history of medication or other allergy that contraindicates their participation
* Use of prescription or non-prescription medications
* History of excessive alcohol use
* History of drug abuse within 6 months of screening
* Use of any illegal drug within 30 days of screening and throughout participation in the study
* History of smoking or use of nicotine containing products within 3 months of screening and throughout participation in the study
* Donation of blood or plasma 4 weeks prior to dosing
* Participation in a clinical trial and has received medication within 30 days
* Weight <50 kg or BMI outside range of 18-32 kg/m2
* Positive for HIV antibody, hepatitis B virus surface antigen, or hepatitis C virus
* Unwillingness to abstain from sexual intercourse with a pregnant or lactating woman and, if engaging in sexual intercourse with a female partner of child-bearing potential, use a condom and spermicide, in addition to having their female partner use another form of contraception, and abstain from sperm donation

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the maximum observed plasma concentration (Cmax) | 9-days
Evaluate the time at which the maximum plasma concentration was observed (tmax) | 9-days
Evaluate the area under the plasma concentration-time curve from time 0 to the last measurable plasma concentration (AUC0-t) | 9-days
Evaluate the area under the plasma concentration-time curve from time 0 to time extrapolated to infinity (AUC0-inf) | 9-days
Evaluate the apparent elimination half-life (t1/2) | 9-days
Evaluate the apparent clearance (CL/F) | 9-days

SECONDARY OUTCOMES:
Safety and tolerability as measured by adverse events | 9-days
Safety and tolerability as measured by clinical observations | 9-days
Safety and tolerability as measured by 12-lead ECGs | 9-days
Safety and tolerability as measured by cardiac telemetry monitoring | 9-days
Safety and tolerability as measured by vital signs (BP, HR, RR and oral temperature) | 9-days
Safety and tolerability as measured by oxygen saturation | 9-days
Safety and tolerability as measured by safety laboratory tests | 9-days

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio, Texas, United States